CLINICAL TRIAL: NCT04994431
Title: Post-Operative Urinary Retention (POUR) in Thoracic Surgery Patients Receiving Prophylactic Tamsulosin
Acronym: POUR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: inability to recruit
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: UMass Memorial Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00018178
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Thoracic Diseases; Urinary Retention
MeSH Terms: conditions — Thoracic Diseases; Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: All subjects that sign a study consent and meet inclusion and exclusion criteria will receive the the study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative Tamsulosin Hydrochloride (Experimental): Participants undergoing thoracic surgery will receive 0.4mgTamsulosin Hydrochloride orally nightly for the two nights immediately prior to surgery and the morning of surgery.
  Interventions: Drug: Tamsulosin Hydrochloride
- Historical Comparator (No Intervention): Participants who underwent thoracic surgery (historical). Information about occurrence of Peri-Operative Urinary Retention in thoracic surgery patients will be obtained via retrospective chart review.

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride — 0.4mg orally nightly for the two days immediately prior to surgery and the morning of surgery.
  Arms: Perioperative Tamsulosin Hydrochloride

SUMMARY:
Post-Operative Urinary Retention (POUR) in Thoracic Surgery is a prospective interventional study aiming to test the hypothesis that the prophylactic use of tamsulosin prior to thoracic surgery in high risk patients leads to reduce the rates of POUR.

DETAILED DESCRIPTION:
Post-operative urinary retention (POUR) is one of the most common post-operative complications encountered by most surgical specialties. The incidence of POUR can vary from five to 70%.

Post-operative urinary retention is a prevalent complication. Patients who undergo thoracic surgery have greater urinary retention rates compared to others. Data on effective methods to reduce the risk of POUR in this high-risk group are limited.

All subjects who meet inclusion and exclusion criteria will be invited to participate. There will be no randomization. All will receive tamsulosin in the pre operative period.

ELIGIBILITY:
Inclusion Criteria:

* All male patients >=60 years old who undergo inpatient thoracic surgery for major resections.

Exclusion Criteria:

* - Prisoners
* Adults unable to consent
* End stage renal disease on hemodialysis
* Indwelling urinary catheter
* Child-Pugh class C hepatic failure
* Usage of the following medications prior to surgery: strong CYP 3A4 inhibitors, strong CYP2D6 inhibitors, other alpha-adrenergic blocking agents, PDE5 inhibitors, and cimetidine
* patients known to be CYP2D6 poor metabolizers
* History of prostatectomy or cystectomy
* Patients with contraindications to tamsulosin and those at high risk for side effects: hypersensitivity to tamsulosin HCl or any component of FLOMAX capsules, hypersensitivity to sulfonamides. History of known glaucoma, hypotension, plan to undergo cataract surgery in the next 2 weeks

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feiran Lou, MD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Memorial Healthcare, Inc., Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Perioperative Tamsulosin Hydrochloride | Historical Comparator
Started | 8 | 101
Completed | 7 | 101
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perioperative Tamsulosin Hydrochloride | Historical Comparator | Total
Number analyzed (Participants) | 7 | 101 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 27 | 29
  >=65 years | 5 | 74 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8) | 70 (7) | 70 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 101 | 108
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 101 | 108

OUTCOME MEASURES:

1. Primary Outcome: Participants With Post-Operative Urinary Retention (Pour)
Description: Proportion of Participants experiencing Post-Operative Urinary Retention (POUR) following thoracic surgery as compared to historic controls.
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Perioperative Tamsulosin Hydrochloride | Historical Comparator
Number analyzed (Participants) | 7 | 101
participants | 1 | 32

ADVERSE EVENTS:
Time Frame: 5 Days
Arm/Group | Perioperative Tamsulosin Hydrochloride | Historical Comparator
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/101
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/101
Other Adverse Events (participants affected / at risk) | 0/7 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perioperative Tamsulosin Hydrochloride (N=7) | Historical Comparator (N=101)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Aspiration requiring intubation

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Difficulty with recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04994431/Prot_SAP_001.pdf